CLINICAL TRIAL: NCT03426878
Title: Exome Sequencing in Diverse Populations in Colorado & Oregon
Brief Title: Cancer Health Assessments Reaching Many
Acronym: CHARM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH); University of Washington (Other); Seattle Children's Hospital (Other); University of California, San Francisco (Other); Denver Health and Hospital Authority (Other); Emory University (Other); Dana-Farber Cancer Institute (Other); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2U01HG007292-05 (NIH); 2U01HG007292-05 (NIH)
Record Dates: First submitted 2018-01-11; First posted 2018-02-08 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-03

CONDITIONS: Hereditary Cancer Syndrome
Keywords: Lynch syndrome; Hereditary breast and ovarian cancer
MeSH Terms: conditions — Neoplastic Syndromes, Hereditary; Colorectal Neoplasms, Hereditary Nonpolyposis; Hereditary Breast and Ovarian Cancer Syndrome

STUDY DESIGN:
Intervention Model Description: All participants will receive exome sequencing. The randomization will be into one of two types of genetic counseling - traditional and modified.
Who Masked: Participant
Masking Description: The participant will not know if they are receiving traditional or modified genetic counseling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional genetic counseling (Active Comparator): This will be typical genetic counseling that a patient would receive in a traditional genetic counseling setting.
  Interventions: Other: Traditional genetic counseling
- Modified genetic counseling (Experimental): This will be genetic counseling that is modified for a lower literacy patient and will include fewer technical terms and less complicated genetic information.
  Interventions: Other: Modified genetic counseling

INTERVENTIONS:
Other: Modified genetic counseling — After participants at high risk for a hereditary cancer syndrome receive exome sequencing, they will receive modified genetic counseling to help them understand the results.
  Arms: Modified genetic counseling
Other: Traditional genetic counseling — After participants at high risk for a hereditary cancer syndrome receive exome sequencing, they will receive traditional genetic counseling to help them understand the results.
  Arms: Traditional genetic counseling

SUMMARY:
The CHARM (Cancer Health Assessment Reaching Many) study will assess the utility of clinical exome sequencing and how it affects care in diverse populations. The study population includes adults at risk for hereditary cancer syndromes.

The primary objective is to implement a hereditary cancer risk assessment program in healthy 18-49 year-olds in primary care settings within a vertically integrated health delivery system (Kaiser Permanente) and a federal qualified health center (Denver Health). The investigators will assess clinical exome sequencing implementation and interpretation, as well as tailored interactions for low health literacy including a contextualized consent process, and a modified approach to results disclosure and genetic counseling. The investigators will also assess the clinical utility (healthcare utilization and adherence to recommended care) and personal utility of primary and additional results from clinical exome sequencing, and evaluate the ethical and policy implications of considering personal utility of genomic information decisions for health care coverage.

DETAILED DESCRIPTION:
Aim 1. Implement a hereditary cancer risk-assessment program in healthy 18-49-year-old adults in primary care settings, with stakeholder input, and offer exome sequencing to clarify risk.

Aim 1A. Identify and recruit 880 adult participants at-risk of a hereditary cancer syndrome.

Aim 1B: Generate medical exome sequence data and interpret variants. Aim 1C: Disclose findings from medical exome sequencing, incorporate results into the electronic medical record (EMR), and facilitate downstream patient management and coordination of care with the provider.

Aim 1D. Engage stakeholders to tailor and optimize the program in diverse populations.

Aim 2. Evaluate and tailor for diverse populations the critical interactions in the program, including the consent process, choices for reporting additional findings, and the response to results disclosure.

Aim 2A. Design, implement, and assess a contextualized consent process to support informed decision-making about participation in research about medical exome sequencing.

Aim 2B. Design, implement, and compare a novel decision aid in the second half of the study for selecting the optional categories of additional findings with the approach we developed in CSER1 that offered a category checklist.

Aim 2C. Design, implement, and compare a modified (communication-focused) approach to results disclosure, genetic counseling, and decision making with a standard (information-focused) approach.

Aim 3. Evaluate the clinical utility (including personal utility) of using exome sequencing to diagnose individuals with hereditary cancer syndromes and provide additional findings.

Aim 3A: Measure the yield of reportable findings for hereditary cancer syndromes and additional findings.

Aim 3B: Evaluate subsequent healthcare utilization for all study participants and adherence to recommended care among individuals who are identified with a hereditary cancer syndrome in diverse settings.

Aim 3C. Assess the personal utility of exome sequencing, including primary and additional findings.

Aim 4. Address pragmatic and ethical challenges to the integration of genomic medicine into clinical and health systems decision-making.

Aim 4A: Develop and pilot a system that integrates genomic, clinical, and healthcare utilization data to inform clinicians and patients acting on genomic information and to reduce care gaps in patient management.

Aim 4B: Advance the analysis of the ethical and policy implications of incorporating personal utility of genomic information into the decision framework for healthcare coverage.

ELIGIBILITY:
Inclusion Criteria:

* Kaiser Permanente Northwest or Denver Health patient
* Screens as high risk for a hereditary cancer syndrome via the risk assessment tool algorithms OR have unknown family history on either their mother or father's side of the family (or both)
* No known prior testing for familial mutations predisposing them to Lynch syndrome or hereditary breast and ovarian cancer
* English or Spanish speaker

Exclusion Criteria:

* Participant self-reported prior testing for Lynch syndrome (LS) or Hereditary Breast and Ovarian Cancer (HBOC) syndrome or identified as having previous comprehensive testing via Kaiser Permanente data files
* Not an English or Spanish speaker
* Unable to provide informed consent
* Don't want results placed in their medical record

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 967 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Leo, PhD, Principal Investigator — Center for Health Research, Kaiser Permanente Northwest; Benjamin S Wilfond, MD, Principal Investigator — Seattle Children's Hospital
Locations (2):
- United States (2):
  - Denver Health, Denver, Colorado
  - Kaiser Permanente Center for Health Research, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Genotype and Phenotype data will be uploaded to ANVIL. Variant data will be uploaded to ClinVar.
Time Frame: Data will be loaded to ANVIL and ClinVar at least annually beginning in 2018.
Access Criteria: Subject to ANVIL and ClinVar regulations.
URL: https://www.genome.gov/Funded-Programs-Projects/Computational-Genomics-and-Data-Science-Program/Genomic-Analysis-Visualization-Informatics-Lab-space-AnVIL

REFERENCES:
- [Derived] Okuyama S, White LL, Anderson KP, Medina E, Deutsch S, Ransom C, Jackson P, Kauffman TL, Mittendorf KF, Leo MC, Bulkley JE, Wilfond BS, Goddard KA, Feigelson HS. Evaluating cancer genetic services in a safety net system: overcoming barriers for a lasting impact beyond the CHARM research project. J Community Genet. 2023 Jun;14(3):329-336. doi: 10.1007/s12687-023-00647-x. Epub 2023 May 1. PMID 37126135
- [Derived] Mittendorf KF, Lewis HS, Duenas DM, Eubanks DJ, Gilmore MJ, Goddard KAB, Joseph G, Kauffman TL, Kraft SA, Lindberg NM, Reyes AA, Shuster E, Syngal S, Ukaegbu C, Zepp JM, Wilfond BS, Porter KM. Literacy-adapted, electronic family history assessment for genetics referral in primary care: patient user insights from qualitative interviews. Hered Cancer Clin Pract. 2022 Jun 10;20(1):22. doi: 10.1186/s13053-022-00231-3. PMID 35689290
- [Derived] Mittendorf KF, Kauffman TL, Amendola LM, Anderson KP, Biesecker BB, Dorschner MO, Duenas DM, Eubanks DJ, Feigelson HS, Gilmore MJ, Hunter JE, Joseph G, Kraft SA, Lee SSJ, Leo MC, Liles EG, Lindberg NM, Muessig KR, Okuyama S, Porter KM, Riddle LS, Rolf BA, Rope AF, Zepp JM, Jarvik GP, Wilfond BS, Goddard KAB; CHARM study team. Cancer Health Assessments Reaching Many (CHARM): A clinical trial assessing a multimodal cancer genetics services delivery program and its impact on diverse populations. Contemp Clin Trials. 2021 Jul;106:106432. doi: 10.1016/j.cct.2021.106432. Epub 2021 May 11. PMID 33984519

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between August 2018 and August 2020 through email, text, and post-cards. Interested patients between 18 and 49 years completed a web-based family history risk assessment to determine eligibility. Participants who screened as high risk were provided with the options to receive exome based panel testing through the study. Participants who consented were provided a saliva sample collection kit that could be returned by mail or to their clinic.
Pre-assignment Details: 967 people were eligible and consented. Of those, 827 submitted a sample for testing. 131 of those people were lost to follow up, declined to receive results, or received a mailed letter with their results. Every outcome measure defined a different analytic sample. Randomization was implemented for only one of the study aims and only applies to outcome measures 6 and 7. Randomization occurred after test results were available.
Groups:
- People Were Eligible and Consented: All individuals eligible and consent for the study
Period: Overall Study
Arm/Group | People Were Eligible and Consented
Started (Eligible and consented) | 967
Submitted a Sample for Testing | 827
Total Who Received Results (Total who received results through either "Traditional Genetic Counseling" or "Modified Genetic Counseling") | 696
Received Results in "Traditional Genetic Counseling" Arm | 344
Received Results in "Modified Genetic Counseling" Arm | 352
Completed (Total randomized who completed the post-results survey and were included in analyses.) | 582
Not Completed | 385
Not completed — Did not return saliva sample to laboratory | 126
Not completed — DNA extraction and sequencing was not successful | 14
Not completed — Declined to receive results | 3
Not completed — Received negative results by mailed letter | 65
Not completed — Lost to Follow-up | 177

BASELINE CHARACTERISTICS:
Groups:
- Baseline Participants: All participants who were eligible and consented
Arm/Group | Baseline Participants
Number analyzed (Participants) | 967
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned at birth
  Participants
    Female | 759
    Male | 208
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian, non-Hispanic | 53
  Black or African American, non-Hispanic | 57
  Hispanic/Latino(a) | 337
  White or European American, non-Hispanic | 438
  Selected multiple racial categories, non-Hispanic | 47
  Selected another racial category | 28
  Unknown | 7
Household income [Count of Participants; unit: Participants]
  Less than $60,000 per year | 489
  $60,000 to less than $100,000 per year | 200
  $100,000 or greater per year | 141
  Unknown/missing | 137
Education level [Count of Participants; unit: Participants]
  Less than high school graduate | 103
  High school graduate or equivalent | 89
  Some post-high school training | 186
  Associate (2-year) college or occupational, technical, or vocational program degree | 123
  Bachelor's degree (for example: BA, AB, BS) | 201
  Graduate or professional degree (for example: MA, MBA, JD, MD, PhD) | 136
  Unknown/missing | 129

OUTCOME MEASURES:

1. Primary Outcome: Positive Findings for Hereditary Cancer Syndromes
Description: Number of people found to have a pathogenic (P) or likely pathogenic (LP) variant in one of the cancer genes associated with Lynch syndrome or hereditary breast and ovarian cancer
Time Frame: For each person, the test result was available within approximately one month of the receipt of that person's specimen at the laboratory.
Population: CHARM participants who were sent a saliva collection kit, returned their sample to the laboratory, had successful DNA extraction, and sequencing was completed. There was no randomization, and therefore no separate "arms" for this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Participants With a Viable Sample: CHARM participants who were sent a saliva collection kit, returned their sample to the laboratory, had successful DNA extraction, and sequencing was completed.
Arm/Group | Participants With a Viable Sample
Number analyzed (Participants) | 827
Participants
  P/LP variant associated w breast and/or ovarian cancer risk | 28
  P/LP variant associated with colon cancer risk | 8
  P/LP variant associated with cancer risk but not with breast, ovarian, colon, or endometrial cancer | 4
  No variant associated with cancer risk found | 787

2. Secondary Outcome: Positive Findings for Other Medically Actionable Genetic Conditions
Description: Number of people with pathogenic variants found in genes related to medically actionable hereditary conditions (other than cancer)
Time Frame: as for outcome 1
Population: 827 is the number of CHARM participants who were sent a saliva collection kit, returned their sample to the laboratory, had successful DNA extraction, and sequencing was completed. There was no randomization, and therefore no separate "arms" for this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With a Viable Sample
Number analyzed (Participants) | 827
Participants | 9

3. Secondary Outcome: Positive Findings for a Selected List of Carrier Conditions
Description: Number of people with pathogenic variants found in genes related to common carrier conditions
Time Frame: as for outcome 1
Population: 810 is the number of CHARM participants who were sent a saliva collection kit, returned their sample to the laboratory, had successful DNA extraction, affirmatively chose to receive "additional findings", and sequencing was completed. Samples from participants who did not choose additional findings were not tested for carrier conditions. There was no randomization, and therefore no separate "arms" for this analysis.
  .
Measure: Count of Participants; unit: Participants
Groups:
- Participants Who Consented to "Additional Genetic Findings": CHARM participants who consented to "additional genetic findings".
Arm/Group | Participants Who Consented to "Additional Genetic Findings"
Number analyzed (Participants) | 810
Participants | 55

4. Secondary Outcome: Number of Participants With Healthcare Utilization Measured Via Electronic Medical Record (EMR) Data
Description: Downstream healthcare utilization of specific recommended procedures (e.g., colonoscopy, mammography, surgery) will be compared between CHARM participants who received at least one actionable risk management recommendation from study genetic counselors and those who did not receive an actionable risk management recommendation.
Time Frame: Within 12 months of participant receiving information about their hereditary cancer syndrome risk
Population: For this analysis participants were not pre-specified to be separated by type of genetic counseling administered. The analysis sample excluded participants: 1) inadequate exome sequencing sample; 2) died or disenrolled before result disclosure; 3) for each procedure (e.g. mammography, colonoscopy, risk-reducing mastectomy ) individuals without relevant organ(s) at study entry. 4) Except for colonoscopy, those who did not reported their sex at birth as female.
Measure: Count of Participants; unit: Participants
Groups:
- Participants With an Actionable Risk Management Recommendation: Participants who received at least one actionable risk management recommendation from study genetic counselors
- Participants Without an Actionable Risk Management Recommendation: Participants who did not receive at least one actionable risk management recommendation from study genetic counselors
Arm/Group | Participants With an Actionable Risk Management Recommendation | Participants Without an Actionable Risk Management Recommendation
Number analyzed (Participants) | 12 | 668
Participants | 6 | 153

5. Secondary Outcome: Participant Understanding of Recommended Care
Description: Measurement of participant's understanding of the recommended care based on their genetic test result will be assessed using a validated survey tool
Time Frame: 2 weeks post result disclosure, 6 months post result disclosure
Population: The study determined that collecting the data on this secondary outcome was not feasible and did not include these questions on surveys or interviews. We did not analyze this outcome.
Arm/Group | Traditional Genetic Counseling | Modified Genetic Counseling
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Participant Understanding of Genetic Test Results
Description: "Perceived understanding of results" This novel 5-item measure asked, "Thinking about only your cancer genetic test result, please rate how strongly you agree or disagree with each of the following statements." The 5 items were assessed on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). A principal-axis factor analysis strongly supported a 1 factor solution (accounting for 65.4% of the variance in these items), providing evidence for structural validity, and a Cronbach's α of 0.90, providing strong evidence for internal consistency. The scale was scored using the mean; thus, the possible scores can range from 1 to 5, with higher scores indicating greater understanding.
Time Frame: 2 weeks post genetic result disclosure
Population: Of the 827 patients with samples sequenced, 352 received results using modified genetic counseling and 344 received results using traditional genetic counseling. A total of 65 patients received their negative results by mailed letter, 3 declined to receive results, and 63 were lost to follow up. Of the 696 patients randomized, 582 completed the post-results survey. Of these 582, 571 provided the responses required for inclusion in this analysis.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Traditional Genetic Counseling | Modified Genetic Counseling
Number analyzed (Participants) | 290 | 281
score on a scale | 4.38 [4.31 to 4.44] | 4.42 [4.35 to 4.49]

7. Secondary Outcome: Participant Satisfaction of Genetic Counseling
Description: This novel measure consisted of 4 items adapted from the Patient Assessment of Communication Effectiveness scale, 8 items developed by the consortium related to participants' overall satisfaction with the results and experience of results disclosures, and 6 items that focused on key elements of modified genetic counseling. Items were measured on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Using principal-axis factor analyses using oblique rotation, we found the 3-factor solution (accounting for 62.5% of the variance in the items) to provide adequate simple structure with conceptually meaningful factors and thus, created subscale scores for each set of items (6 loaded on each factor): "genetic counseling relationship score", "communication difficulty score", and "communication ease score". The possible mean scores can range from 1 to 5, with higher scores indicating a better outcome.
Time Frame: 2 weeks post genetic results disclosure
Population: The number analyzed in each row differs from overall number analyzed because some participants did not respond to all questions in the survey resulting in missing data. For each analysis we used all available data.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Traditional Genetic Counseling | Modified Genetic Counseling
Number analyzed (Participants) | 296 | 286
score on a scale
  Communication ease score: number analyzed (Participants) | 288 | 274
  Communication ease score | 4.68 [4.62 to 4.73] | 4.70 [4.64 to 4.75]
  Communication difficulty score: number analyzed (Participants) | 280 | 268
  Communication difficulty score | 1.82 [1.72 to 1.92] | 1.83 [1.74 to 1.92]
  Genetic counseling relationship score: number analyzed (Participants) | 274 | 266
  Genetic counseling relationship score | 4.29 [4.22 to 4.35] | 4.37 [4.32 to 4.43]

8. Secondary Outcome: Family Communication
Description: Measurement of the degree to which participants shared their genetic test results with various family members will be assessed using a validated survey tool
Time Frame: Assessed 6 months post result disclosure
Population: For this analysis, participants were not pre-specified to be separated by type of genetic counseling administered. Survey data from 562 CHARM participants who received genetic test results and completed survey questions on family communication were available for analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Participants Who Received Genetic Test Results and Completed Certain Survey Questions: CHARM participants who received genetic test results and completed survey questions on family communication. This outcome measure does not have a comparison group
Arm/Group | Participants Who Received Genetic Test Results and Completed Certain Survey Questions
Number analyzed (Participants) | 562
Participants | 466

9. Secondary Outcome: Personal Utility of Genomic Sequencing (Qualitative Interview Only)
Description: Participant's perceived utility of obtaining genetic testing and genetic counseling were assessed. Data collection used semi-structured qualitative interviews. Analyses were conducted using a modified grounded theory approach and explored the five utility domains of the model: clinical, emotional, behavioral, cognitive, and social. The analysis examined how well this multifaceted perceived utility model applied to the responses provided during the interviews. The qualitative data was not quantified in any way and can not be represented in a tabular format.
Time Frame: Qualitative interviews were conducted within 1 month of results disclosure; a subset of these participants were interviewed again at 6 months post-results disclosure.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: N/a. Adverse event data was not collected for this study. This data would not result from the CHARM study procedures. The IRB did not require adverse event data collection.
Description: No study-related adverse events would reasonably be expected to result from the CHARM study procedures. The IRB did not require adverse event data collection.
Groups:
- All Enrolled Participants: Participants who enrolled in the CHARM study who were sent a saliva collection kit. There was no randomization, and therefore no separate "arms" for this analysis.
Arm/Group | All Enrolled Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/78/NCT03426878/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/78/NCT03426878/ICF_001.pdf